CLINICAL TRIAL: NCT00835419
Title: An Open Label, Multicentre, Two Stage, Phase II Study To Evaluate Efficacy And Safety Of P276-00 In Subjects Of Malignant Melanoma Positive For Cyclin D1 Expression
Brief Title: Efficacy Study Of P276-00 In Subjects Of Malignant Melanoma Positive For Cyclin D1 Expression
Acronym: ENVER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P276-00/27/08
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Melanoma
Keywords: metastatic malignant melanoma with cyclin D1 positivity
MeSH Terms: conditions — Melanoma | interventions — P276-00

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): P276-00 investigational product (small molecule Cdk 4-D1, Cdk1-B and Cdk9-T inhibitor)
  Interventions: Drug: P276-00

INTERVENTIONS:
Drug: P276-00 — P276-00 -small molecule Cdk 4-D1, Cdk1-B and Cdk9-T inhibitor

SUMMARY:
The purpose of this study is to evaluate efficacy of P276-00 in subjects with advanced malignant melanoma positive for cyclin D1 expression

DETAILED DESCRIPTION:
Currently, melanoma is the fifth most common cancer diagnosed in men and the seventh most common cancer diagnosed in women.Advanced melanoma has a very poor prognosis.For a vast majority of subjects with malignant melanoma, there are no effective therapies.Therefore, the development of effective therapies for this subject population remains a priority in oncology.In a limited study in melanomas, increased cyclin D1 protein expression, as was observed in 33% cases.P276-00 is a novel potent small molecule flavone derived Cyclin dependent kinase (Cdk) Cdk 4-D1, Cdk1-B and Cdk9-T inhibitor.P276-00 demonstrated significant and selective antiproliferative effect against melanoma cell lines.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with histologically confirmed stage III (unresectable) or stage IV metastatic melanoma as per revised AJCC melanoma staging
2. Subject positive for cyclin D1 expression by appropriate technique
3. Subject with at least one metastasis in which surgery was not a curative option and had relapsed from, or had not responded to at least one regimen containing Dacarbazine and or IL-2
4. Subjects with measurable disease [at least one unidimensionally measurable lesion ³ 20 mm with conventional techniques (CT, MRI, X-ray) or ³ 10 mm by spiral CT scan]
5. Subject of either sex and 18 years of age or elder
6. Eastern Cooperative Oncology Group (ECOG) performance status 2 or less
7. Subject with life expectancy of at least 4 months
8. Subject must have normal organ and marrow function as defined below

   * Hemoglobin ≥ 9 g/dL
   * Absolute Neutrophil count ≥ 1,500/mm3
   * Platelets ≥ 100,000/mm3
   * Total bilirubin ≤ 1.5 X institutional upper limit of normal (ULN)
   * AST/ALT ≤ 2.5 X institutional ULN or ≤ 5 X ULN if liver function abnormalities are due to underlying malignancy
   * S. creatinine within 1.5 times the upper normal institutional limits
9. Subjects with metastatic disease to the central nervous system will be included provided they had either:

   * No evidence of leptomeningeal disease
   * Resected CNS metastasis without evidence of recurrence for 12 week or more
   * Brain metastasis treated by radiosurgery without evidence of recurrence or progression for 12 week or more
   * Multiple brain lesions treated with whole brain radiation therapy (WBRT) with stable disease off corticosteroids for 12 week or more prior to start of therapy
10. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Treatment with P276?00 or other cyclin dependent kinase (CDK) targeting agents anytime in the past
2. History of allergic reactions attributed to compounds of chemical composition similar to P276?00
3. Subject who have had chemotherapy, immunotherapy or radiotherapy within 4 week prior to first dosing of study agent. For nitrosoureas, there shall be interval of at least six week from first dosing of study agent
4. Subject who have not recovered from adverse events (AE ³ CTCAE Grade 2) due to agents administered more than 4 week earlier.
5. Subject who had received any other investigational drug within 1 month prior to day 1 of study drug administration
6. Prior malignancy (within the last 3 years) except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, in situ prostate cancer or any other cancer for which the subject has been disease-free for at least 3 years
7. Any medical condition (such as but not limited to severe/unstable angina, history of myocardial infarction, coronary/peripheral artery bypass graft, symptomatic congestive cardiac failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism) or laboratory abnormality(ies) which might make it difficult for the subject to participate in the study, at the discretion of the Principal Investigator (PI)or co-PI
8. Known human immunodeficiency virus (HIV) positivity or acquired immunodeficiency syndrome (AIDS) related illness
9. QTc > 470 millisecond on 12 lead Electrocardiogram at screening
10. Pregnant or nursing women
11. Women of childbearing potential [defined as a sexually mature woman who has not undergone hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e. who has had menses any time in the preceding 24 consecutive months)] and men, not agreeing to use adequate contraception (e.g., hormonal or barrier method of birth control or abstinence) after signing an informed consent document (ICD), during the duration of study participation and for at least 4 week after withdrawal from the study, unless they are surgically sterilized

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-05; Primary Completion 2011-04 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival rate at Day 168 | 168 days

SECONDARY OUTCOMES:
Overall survival rate at 1 year, objective response rate,duration of response | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hersey, MD, Principal Investigator — Newcastle University
Locations (7):
- Australia (4):
  - University of Newcastle, School of Medicine and Public Health, Newcastle, New South Wales
  - Mater Adult Hospital Raymond Tce South Brisbane, QLD 4101, Brisbane
  - Peninsula Oncology Centre, Frankston
  - John Fawkner Cancer Trial Centre, Victoria
- India (2):
  - Curie Manavata Cancer Center, Nashik, Maharashtra
  - Chhatrapati Shahuji Maharaj Medical University, Lucknow, Uttar Pradesh
- Christchurch Oncology Research Unit, Oncology Service, Christchurch Hospital, Riccarton Avenue, Private Bag 4710, Christchurch,, Christchurch, New Zealand